CLINICAL TRIAL: NCT06144359
Title: Role of Diffusion Tensor Brain MRI in the Detection of Structural Abnormality of the Apparently Normal White Substance in Patients Victims of Concussion in the Context of Sport : Prospective Comprative Study Versus Healthy Subjects
Brief Title: Diffusion Tensor Brain MRI in the Detection of Structural Abnormality of the White Substance in Concussion
Acronym: COMMOTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2022 CLAISE
Record Dates: First submitted 2023-10-05; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Concussion, Brain
Keywords: concussion; diffusion tensor imaging; 3 Teslas; sport
MeSH Terms: conditions — Brain Concussion | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concussed patients (Experimental): Patients will be included :
  * Sports patients with concussion in sport,
  * Consultation with Sports Medecine within 7 days of concussion.
  * affiliated to a social security scheme.
  Interventions: Other: specific MRI Acquisition (Diffusion Tensor Imaging) at 3T
- Control subjects (Experimental): * major case matched subjects by sex and age (± 5 years).
  * affiliated to a social security scheme.
  * written consent.
  Interventions: Other: specific MRI Acquisition (Diffusion Tensor Imaging) at 3T

INTERVENTIONS:
Other: specific MRI Acquisition (Diffusion Tensor Imaging) at 3T — The imaging will be carried out on the technical stage of the 3T MRI Research of the University Hospital of Clermont-Ferrand with the following sequences:
  - For traumatized and healthy subjects: MRI 3 Teslas (3D T1, T2 axial TSE, T2* axial, SWI axial, Sagittale cube FLAIR, DTI 20-direction sequence) The image processing will be carried out within the radiology department: morphological analysis and analysis of tractography and diffusion parameters (FA and ADC, diffusivity) on predefined and reproducible Regions of Interest (ROIs).
  Regions Of Interest include: splenium of the corpus callosum, internal capsule, cortico-spinal tract, optic radiation.

SUMMARY:
Concussions in sports are a major public health problem because of their frequency, and are often underdiagnosed because of an unspecific clinical picture or sometimes masked by the concussion itself.

Support data has been constantly evolving in recent years, including the last publication of the Berlin Consensus in 2016 specifying support in the field. However, to date, there is no tool to predict the severity of a concussion or to predict when it will return to play objectively and reliably.

Brain MRI done after the head injury is most often normal. However, previous studies agree that there is a persistent electrophysiologic disturbance several weeks after the injury, and the specific pathophysiology of white matter changes after a head injury remains controversial.

Diffusion tensor imaging (DTI), in addition to morphological sequences, is capable of assessing white matter microstructure and fibrous tract integrity or not. Several parameters, such as the seemingly normal white matter fractional anisotropy (FA) coefficient, the mean diffusivity and the radial diffusivity, may be altered in the aftermath of a concussion, indicating axonal damage not visible on conventional MRI sequences.

Previous studies have evaluated these parameters with sometimes contradictory results: some have found an increase in AF in specific regions such as the cortico-spinal tract and the corpus callosum, others have found a decrease in AF.

So far, assessment of a player's condition on and off the field after a head injury has been based on clinical criteria alone, sometimes far too subjective. The player may choose to mask their symptoms to allow them to return to the game faster, or feign more than they have. Once pathologies such as bone fractures or intracranial hematomas are ruled out by conventional imaging, there is no longer any tool for a more accurate diagnosis of possible microstructural alterations of brain tissue and for monitoring of the patient.

The advent of new MRI techniques such as diffusion imaging, and particularly diffusion tensor imaging (DTI), is a promising tool to better understand white matter involvement in diffuse axonal lesions.

DETAILED DESCRIPTION:
Diffusion imaging is based on analyzing the movements of water molecules in a tissue. The parameter measuring the intensity of this diffusion is the apparent coefficient of diffusion (ADC) which varies in particular as a function of the cell density. Diffusion imaging is therefore a modality that reflects tissue density, and in this case is capable of revealing pathological processes in white matter.

Diffusion tensor imaging (DTI), a newer and complementary modality, allows estimation of the preferred directions of diffusion of water molecules in a tissue.

Compared to "single" scattering imaging that uses scattering gradients applied in 3 directions, DTI uses these same gradients applied in at least 6 directions (20 for our study).

In white matter, diffusion is constrained by the axon cell membrane and the myelin sheath, and preferably follows the fiber bundles tangentially. Diffusion tensor modeling allows the determination within a voxel of the principal direction (maximum diffusivity) of proton motion, which corresponds to the orientation of the white matter fibers.

Thus, DTI allows the study of tissue microstructural organization. This degree of organization of SB is measurable through diffusion tensor parameters, such as the fraction of anisotropy or fractional anisotropy (FA). When the diffusion is constrained in a main direction, it is said to be anisotropic and the FA tends towards 1. On the other hand, when it is carried out indifferently in all directions of space, it is said to be isotropic and the FA then tends towards a zero value.

It would appear, therefore, that DTI may be a more sensitive means than diffusion for revealing apparently normal SB abnormalities related to head trauma

For patients who have a concussion, doctors in the sports medicine department will offer them MRI after the visit. At this visit, the investigator will inform (orally and in writing) the subject about the study and, after obtaining the subject's consent, note demographic and clinical information, date of concussion, complications, medical history and SCAT 5 (standardized tool for concussions) score. After the inclusion and exclusion criteria have been verified, the participant will be invited within 7 days to perform an MRI.

For control subjects, following presentation of the study by one of the investigators, they will be summoned for the baseline visit followed by the first MRI. The 15-minute baseline visit will be conducted by one of the study investigators. The investigator will inform (orally and in writing) the subject about the study and after obtaining their consent will record demographic information, medical history and check inclusion and exclusion criteria. MRI will be done next.

After a delay of 1 month ± 5 days, the second MRI will be scheduled for all subjects.

The first MRI consists of several sequences (the total acquisition time is less than one hour) (no contrast injection for these tests). The second is shorter and involves the acquisition of the sequence in diffusion voltage (7 minutes) and that of anatomical locating images (4 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Cases: Sports patients with concussion in sport, seen in Sports Medicine consultation within 7 days of concussion.
* Healthy controls: major case matched subjects by sex and age (± 5 years).
* For all: people with health insurance

Exclusion Criteria:

* For all: major minor or incapacitated people, with a history of neurological or psychiatric disease, people who have had concussions in the past, pregnant or breastfeeding women, protected persons (guardianship, curatorship, safeguard of justice), contraindication to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
White matter microstructure lesions on DTI sequence | MRI at Day 0, Day 30 and comparison intra- and inter-group
  Number of participants with white matter microstructure lesions on DTI sequence on IRM at Day 0 and Day 30

SECONDARY OUTCOMES:
Tractography parameters measured in splenium of the corpus callosum, internal capsule, cortico-spinal tract, optic radiation. | Measurement at MRI at Day 0, Day 30 and comparison intra- and inter-group
  Measurement of FA (fraction of anisotropy) after ROI is applied in the regions of the brain studied and then intra-group and inter-group comparison.
  Regions Of Interest include: splenium of the corpus callosum, internal capsule, cortico-spinal tract, optic radiation.
Tractography parameters measured in splenium of the corpus callosum, internal capsule, cortico-spinal tract, optic radiation. | Measurement at MRI at Day 0, Day 30 and comparison intra- and inter-group
  Measurement of diffusion parameters (axial, radial diffusion) after ROI is applied in the regions of the brain studied and then intra-group and inter-group comparison.
  Regions Of Interest include: splenium of the corpus callosum, internal capsule, cortico-spinal tract, optic radiation.
Tractography parameters measured in splenium of the corpus callosum, internal capsule, cortico-spinal tract, optic radiation. | Measurement at MRI at Day 0, Day 30 and comparison intra- and inter-group
  Measurement of ADC (apparent coefficient of diffusion) tractography parameters after ROI is applied in the regions of the brain studied and then intra-group and inter-group comparison.
  Regions Of Interest include: splenium of the corpus callosum, internal capsule, cortico-spinal tract, optic radiation.
Relationships between white matter microstructure lesion and physical examination in Sports medicine | Sports medicine within 7 days after concussion
  Investigate the relationships between these abnormalities (damage to white matter microstructure apparently normal on classical sequences) to the physical examination in Sports medicine using the Sport Concussion Assessment Tool 5th Edition scale.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clemront-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavlovic D, Pekic S, Stojanovic M, Popovic V. Traumatic brain injury: neuropathological, neurocognitive and neurobehavioral sequelae. Pituitary. 2019 Jun;22(3):270-282. doi: 10.1007/s11102-019-00957-9. PMID 30929221
- [Result] Cubon VA, Putukian M, Boyer C, Dettwiler A. A diffusion tensor imaging study on the white matter skeleton in individuals with sports-related concussion. J Neurotrauma. 2011 Feb;28(2):189-201. doi: 10.1089/neu.2010.1430. Epub 2011 Jan 27. PMID 21083414
- [Result] Lancaster MA, Meier TB, Olson DV, McCrea MA, Nelson LD, Muftuler LT. Chronic differences in white matter integrity following sport-related concussion as measured by diffusion MRI: 6-Month follow-up. Hum Brain Mapp. 2018 Nov;39(11):4276-4289. doi: 10.1002/hbm.24245. Epub 2018 Jul 2. PMID 29964356
- [Result] Chappell MH, Ulug AM, Zhang L, Heitger MH, Jordan BD, Zimmerman RD, Watts R. Distribution of microstructural damage in the brains of professional boxers: a diffusion MRI study. J Magn Reson Imaging. 2006 Sep;24(3):537-42. doi: 10.1002/jmri.20656. PMID 16878306
- [Result] Yin B, Li DD, Huang H, Gu CH, Bai GH, Hu LX, Zhuang JF, Zhang M. Longitudinal Changes in Diffusion Tensor Imaging Following Mild Traumatic Brain Injury and Correlation With Outcome. Front Neural Circuits. 2019 May 7;13:28. doi: 10.3389/fncir.2019.00028. eCollection 2019. PMID 31133818
- [Result] Meier TB, Bergamino M, Bellgowan PS, Teague TK, Ling JM, Jeromin A, Mayer AR. Longitudinal assessment of white matter abnormalities following sports-related concussion. Hum Brain Mapp. 2016 Feb;37(2):833-45. doi: 10.1002/hbm.23072. Epub 2015 Dec 10. PMID 26663463
- [Result] Jang SH, Seo YS. Diffusion tensor tractography characteristics of axonal injury in concussion/mild traumatic brain injury. Neural Regen Res. 2022 May;17(5):978-982. doi: 10.4103/1673-5374.324825. PMID 34558511
- [Result] Gonzalez AC, Kim M, Keser Z, Ibrahim L, Singh SK, Ahmad MJ, Hasan O, Kamali A, Hasan KM, Schulz PE. Diffusion Tensor Imaging Correlates of Concussion Related Cognitive Impairment. Front Neurol. 2021 May 24;12:639179. doi: 10.3389/fneur.2021.639179. eCollection 2021. PMID 34108926